CLINICAL TRIAL: NCT01487707
Title: Strengthening the Midwife Service Scheme With Community Focused Interventions: Evidence From a Randomized Controlled Field Trial in Nigeria
Brief Title: Community Based Strategies to Reduce Maternal Mortality in Northern Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abdul Latif Jameel Poverty Action Lab (Other)
Collaborators: Planned Parenthood Federation Nigeria (Unknown); MacArthur Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 019368-001
Record Dates: First submitted 2011-12-06; First posted 2011-12-07 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Maternal Mortality
Keywords: pregnancy; maternal mortality; neonatal mortality; community intervention; voluntary health worker; safe birth kit; maternal child health
MeSH Terms: conditions — Maternal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Voluntary Health Worker (VHW) Program (Experimental)
  Interventions: Behavioral: Voluntary Health Worker (VHW) Program
- VHW program plus Safe Birth Kit (Experimental)
  Interventions: Behavioral: Voluntary Health Worker (VHW) Program; Behavioral: Safe Birth Kit
- VHW program plus Folk Media Activities (Experimental)
  Interventions: Behavioral: Voluntary Health Worker (VHW) Program; Behavioral: Community Folk Media Campaigns

INTERVENTIONS:
Behavioral: Voluntary Health Worker (VHW) Program — Voluntary Health Workers will conduct door-to-door campaigns on maternal and child health, and will visit pregnant women regularly to to educate and to encourage use of antenatal care and facility-based deliveries.
Behavioral: Safe Birth Kit — A safe birth kit, containing sterile materials to diminish infection risk will be given to pregnant women.
  Arms: VHW program plus Safe Birth Kit
Behavioral: Community Folk Media Campaigns — Community-wide media activities, including dramas, intended to address community norms regarding maternal and child health.
  Arms: VHW program plus Folk Media Activities

SUMMARY:
The objective of this cluster randomized controlled trial is to assess the impact of several community-based interventions that address the key factors underlying the high maternal mortality, as well as neonatal mortality and morbidity in northern Nigeria. The interventions, include:

1. a Voluntary Health Worker Program (VHW)
2. the VHW program with provision of a safe birth kit
3. the VHW program with community folk media activities.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age who live in the study clusters who provide consent.

Exclusion Criteria:

* Eligible women who do not consent.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7200 (Actual)
Dates: Start 2011-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Maternal Mortality Ratio | 42 days post delivery

SECONDARY OUTCOMES:
Maternal Morbidity Rates | 42 days post delivery
Proportion of women delivering in a health facility | 2 years
Neonatal Mortality Rate | 28 days after birth
Proportion of women receiving antenatal care during pregnancy | 2 years
Knowledge of warning signs during pregnancy | 2 years
Proportion of women/newborns receiving postnatal care | 2 years
Birthweight | 2 years
Stunting, underweight and wasting in children under 5 years | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Leight, PhD, Principal Investigator — Massachusetts Institute of Technology; Vandana Sharma, MD, Principal Investigator — Massachusetts Institute of Technology; Martina Bjorkman-Nyqvist, PhD, Principal Investigator — Stockholm School of Economics
Locations (1):
- Planned Parenthood Federation, Abuja, Nigeria

REFERENCES:
- [Derived] Sharma V, Leight J, AbdulAziz F, Giroux N, Nyqvist MB. Illness recognition, decision-making, and care-seeking for maternal and newborn complications: a qualitative study in Jigawa State, Northern Nigeria. J Health Popul Nutr. 2017 Dec 21;36(Suppl 1):46. doi: 10.1186/s41043-017-0124-y. PMID 29297412
- [Derived] Sharma V, Brown W, Kainuwa MA, Leight J, Nyqvist MB. High maternal mortality in Jigawa State, Northern Nigeria estimated using the sisterhood method. BMC Pregnancy Childbirth. 2017 Jun 2;17(1):163. doi: 10.1186/s12884-017-1341-5. PMID 28577546